CLINICAL TRIAL: NCT01980420
Title: Prospective Study of the Impact of Sleeve Gastrectomy on Gastro-esophageal Junction Function
Acronym: FFSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IHU Strasbourg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-001; 2013-A00723-42 (Other: ANSM France)
Record Dates: First submitted 2013-10-28; First posted 2013-11-11 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-08

CONDITIONS: Morbid Obesity
Keywords: Sleeve gastrectomy; Oesogastric junction - GEJ; Dynamic MRI Imaging
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sleeve gastrectomy (Other): All patients will undergo sleeve gastrectomy
  Interventions: Procedure: Laparoscopic sleeve gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic sleeve gastrectomy — Conventional laparoscopic sleeve gastrectomy using EndoFLIP® probe to provide measures on the distensibility of gastro-esophageal junction (GEJ) and gastric tube.

SUMMARY:
Improved results for sleeve gastrectomy could be possible if more was known about the surgical / mechanical factors that affect outcome.

DETAILED DESCRIPTION:
Effectiveness of sleeve gastrectomy is between gastric banding and gastric bypass. However, a proportion of patients that undergo surgery, report troublesome and persistent dysphagia, pain, new onset or worsening of gastro-esophageal reflux (GER) requiring treatment. Improved results for sleeve gastrectomy could be possible if more was known about the surgical / mechanical factors that affect outcome. Current investigations based on traditional intra-luminal imaging (endoscopy) and radiology (UGI series) may not provide adequate preoperative assessment of esophago-gastric dynamics. Current practice in the creation of a sleeve gastrectomy involves the use of a bougie or endoscope around which the sleeve is stapled. There is no consensus on the diameter of this bougie and this intraoperative calibration may alter the gastro-esophageal junction (GEJ) anatomy, does not provide real time physiology feedback, and allows only for a rough approximation of the size of the sleeve providing no information about the distensibility and pressure gradient of the newly created gastric tube as it is filled. A more distensible sleeve will have lower intra-gastric pressure, and thus will theoretically be expected to reduce the incidence of side effects. As laparoscopic sleeve gastrectomy is performed with increasing frequency, there is a need for development of tools to assist the surgeon in modeling properly and standardize the gastroplasty. This study will be based on a strict assessment of the anatomical and functional characteristics of the "ideal "gastric sleeve, using existing imaging modalities (endoscopy - CT scan- MRI - HRM).

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female over 18 years old
* Patient scheduled to undergo a sleeve gastrectomy for obesity
* Patient with surgical indication validated by the obesity multidisciplinary meeting (RCP)
* Patient able to understand the study and to provide written informed consent
* Patient registered with the French social security regime

Non-inclusion criteria:

* Patient unable to give written informed consent
* Patient presenting contra-indication to the conduct of an MRI (claustrophobia, implantable medical devices)
* Patient presenting risks of allergic reaction to MRI contrast agents (gadolinium)
* Patient presenting, in the investigator's judgment, a condition or disease preventing their participation to study procedures
* Patient pregnant or breast-feeding
* Patient within exclusion period from other clinical trial
* Patient having forfeited their freedom of an administrative or legal obligation
* Patient being under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of patients with postoperative GIQLI score greater than preoperative score | 50% excess weight loss (about 6 months post surgery)
  Patients with postoperative GIQLI (Gastro-Intestinal Quality of Life Index) score greater than preoperative score

SECONDARY OUTCOMES:
Quality of life (GIQLI) | 50% of excess weight loss (about 6 months post surgery)
  Quality of life (Gastro-Intestinal Quality of Life Index)
GERD and dysphagia symptoms (GSAS questionnaire) | 50% of excess weight loss (about 6 months post surgery)
  GERD (Gastroesophageal Reflux Disease) Symptom Assessment Scale
Functional examinations | 50% of excess weight loss (about 6 months post surgery)
  Include:
  * Dynamic MRI
  * High resolution manometry
  * pH impedance
  * upper gastro-intestinal study (UGI)
EndoFLIP® measures | Intra-operatively
  Measurements provided by EndoFlip probe : GEJ distensibility, diameter, pressure
Surgical video analysis | within 6 months post surgery
  Analysis of surgery videos to detect technical "errors" explaining clinical and/or functional outcome
Per and post-operative complications | within 6 months post surgery
  Complications occuring during surgery and within 6 months of surgery (reach of 50% of excess weight loss)
Cost of exploratory exams | 50% excess weight loss (about 6 months post surgery)
Cost of exploratory exams | Within 2 months prior to surgery

CONTACTS AND LOCATIONS:
Overall Officials: Silvana Perretta, Pr, Principal Investigator — Service de Chirurgie Digestive et Endocrinienne - Nouvel Hôpital Civil - Strasbourg
Locations (1):
- Service de Chirurgie Digestive et Endocrinienne - Nouvel Hôpital Civil, Strasbourg, France

REFERENCES:
- [Derived] Quero G, Fiorillo C, Dallemagne B, Mascagni P, Curcic J, Fox M, Perretta S. The Causes of Gastroesophageal Reflux after Laparoscopic Sleeve Gastrectomy: Quantitative Assessment of the Structure and Function of the Esophagogastric Junction by Magnetic Resonance Imaging and High-Resolution Manometry. Obes Surg. 2020 Jun;30(6):2108-2117. doi: 10.1007/s11695-020-04438-y. PMID 32207049